CLINICAL TRIAL: NCT03002116
Title: Microwave Radiometry Thermometry for Non-invasive Diagnosis of Arterial Disease in Diabetic Patients With Suspected Critical Limb Ischemia: A Multi-centre Feasibility Study
Brief Title: Microwave Radiometry Thermometry for the Diagnosis of Critical Limb Ischemia in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: University Hospital of Patras (Other); Bolton Research Foundation (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Assistant Professor of Radiology., Attikon Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EBΔ 1310/10-2-16
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Foot; Peripheral Arterial Disease; Ischaemic Neuropathy
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group N (Active Comparator): Healthy volunteers without peripheral arterial disease according to clinical examination and Duplex ultrasound
  Interventions: Other: Tissue thermometry using non-invasive microwave radiometry device
- Group DN (Experimental): Patients suffering from diabetes and diabetic foot without vascular compromise according to clinical assessment continuous-wave Doppler and Duplex ultrasound
  Interventions: Other: Tissue thermometry using non-invasive microwave radiometry device
- Group DC (Experimental): Diabetic patients with Rutherford-Becker 5 or 6 critical limb ischemia, verified by clinical examination, abnormal continuous-wave Doppler or Duplex ultrasound and intra-arterial angiography.
  Interventions: Other: Tissue thermometry using non-invasive microwave radiometry device
- Group NDC (Experimental): Non diabetic patients with Rutherford-Becker 5 or 6 critical limb ischemia, verified by clinical examination, abnormal continuous-wave Doppler or Duplex ultrasound and intra-arterial angiography.
  Interventions: Other: Tissue thermometry using non-invasive microwave radiometry device

INTERVENTIONS:
Other: Tissue thermometry using non-invasive microwave radiometry device — In Patients included in the four study groups underwent non-invasive tissue thermometry using microwave radiometry (MWR) device, at the same room temperature and with the same methodology. Specifically, the probe of the RTM-01-RES (University of Bolton, UK) device was by applied on the surface of the foot tissue at an angle of 90o degrees for approximately 8 to 10 seconds in pre-determined sites. Measurements were performed by two independent operators. Three measurements were taken from each site. The mean value of the three values calculated by the 2 different operators was used for the analysis. Measurements were recorded using a dedicated software.

SUMMARY:
Diagnosis of vascular involvement in diabetic foot disease remains challenging. Differential diagnosis between pure neuropathic or neuro-ischemic diabetic foot requires a combination of clinical examination, medical history and ankle-brachial index (ABI) measurement, which is considered the "gold standard" non-invasive modality for limb ischemia diagnosis. However, in diabetic patients with suspected arterial ischemia resulting in tissue loss (critical limb ischemia; CLI), false negative ABI results are frequent due to Monckeberg medial sclerosis producing incompressible vessels, while clinical signs are subjective and not accurate in posing definite diagnosis of CLI.

The investigators conducted a proof of concept study of the feasibility of microwave radiometry thermometry for non-invasive diagnosis of CLI in diabetic patients with tissue loss.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, trial designed to investigate the he feasibility and efficacy of microwave radiometry thermometry for non-invasive diagnosis of CLI in diabetic patients with tissue loss. The study included 80 patients, equally divided in four groups. Group N: normal subjects; group DN: diabetic patients with verified neuropathic ulcers without vascular involvement; group DC: diabetic patients with CLI and group NDC: non-diabetic patients with CLI. All patients underwent MWR with the RTM -01-RES device (University of Bolton, UK) to record the mean internal tissue temperature of the foot. MWR is based on the principle that the intensity of radiation is proportional to tissue temperature. The specific device is not commercially available and has been developed to detect temperatures from internal tissues at microwave frequencies. Foot temperature measurements were performed as near as possible at the site of ulceration in patients of groups DN, DC and NDC and in various sites in subjects of control group N.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from both insulin and not insulin dependent diabetes mellitus.
* Critical limb ischemia verified by both clinical examination, haemodynamic tests and digital subtraction angiography.

Exclusion Criteria:

* Uncertainty regarding the absence of peripheral arterial disease in groups N and DN.
* Uncertainty regarding the diagnosis of critical limb ischemia for patients in groups DC and NDC.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mean foot tissue temperature | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elias Brountzos, MD, PhD, Study Chair — ATTIKO University General Hospital
Locations (3):
- Greece (2):
  - Patras University Hospital, Rio, Achaia
  - Attiko University General Hospital, Athens, Attica
- Institute for Materials Research and Innovation, University of Bolton, Bolton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided